CLINICAL TRIAL: NCT04248907
Title: Evaluating the Effect of Transtibial Pin Lock Suspension at Varying Distraction Values Using a Modified Air Bladder Casting System
Brief Title: Transtibial Pin Lock Suspension at Varying Distraction Values Using a Modified Air Bladder Casting System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Corona Virus guidelines, we have decided to withdraw the study.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Michael Davidson, Assistant Professor Department of Orthotics and Prothetics, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 5190492
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Amputation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Socket A (Experimental): To eliminate variables while casting the student investigators will be using a system very similar to that of Ossur's ICEX, developed in Reykjavik, Iceland. The ICEX system uses an air bladder system that allows a socket to be constructed directly onto the residuum; resulting in even pressure distribution during the time of casting. The ICEX system will ensure that the student investigators are obtaining consistent socket pressures and that the team will be precisely testing the distraction values on the multiple sockets obtained in this experiment. During this experiment, the researchers will be using a modified air bladder system.
  Interventions: Other: 0 pound tension
- Socket B (Active Comparator): To eliminate variables while casting the student investigators will be using a system very similar to that of Ossur's ICEX, developed in Reykjavik, Iceland. The ICEX system uses an air bladder system that allows a socket to be constructed directly onto the residuum; resulting in even pressure distribution during the time of casting. The ICEX system will ensure that the student investigators are obtaining consistent socket pressures and that the team will be precisely testing the distraction values on the multiple sockets obtained in this experiment. During this experiment, the researchers will be using a modified air bladder system.
  Interventions: Other: 2 pound tension
- Socket C (Active Comparator): To eliminate variables while casting the student investigators will be using a system very similar to that of Ossur's ICEX, developed in Reykjavik, Iceland. The ICEX system uses an air bladder system that allows a socket to be constructed directly onto the residuum; resulting in even pressure distribution during the time of casting. The ICEX system will ensure that the student investigators are obtaining consistent socket pressures and that the team will be precisely testing the distraction values on the multiple sockets obtained in this experiment. During this experiment, the researchers will be using a modified air bladder system.
  Interventions: Other: 4 pound tension

INTERVENTIONS:
Other: 0 pound tension — A digital fish scale will be attached to the distal strap of a gel liner to measure the distraction values while casting. A digital fish scale can measure in pounds or kilograms depending on how you set it. The digital fish scale will be held in place while casting to maintain a consistent tension between the scale and the residual limb.
  Arms: Socket A
Other: 2 pound tension — A digital fish scale will be attached to the distal strap of a gel liner to measure the distraction values while casting. A digital fish scale can measure in pounds or kilograms depending on how you set it. The digital fish scale will be held in place while casting to maintain a consistent tension between the scale and the residual limb.
  Arms: Socket B
Other: 4 pound tension — A digital fish scale will be attached to the distal strap of a gel liner to measure the distraction values while casting. A digital fish scale can measure in pounds or kilograms depending on how you set it. The digital fish scale will be held in place while casting to maintain a consistent tension between the scale and the residual limb.
  Arms: Socket C

SUMMARY:
To assess the effects various distraction values have on the 'slippage' effect of a transtibial pin-lock system

DETAILED DESCRIPTION:
This experiment will consist of a total of four visits. The testing process will consist of a series of castings, surveys, data collection, and outcome testing that includes both endurance and aerobic exercises while wearing the check sockets of varying tension values. The outcome measures will be performed in the Nichol Hall Motion Capture Lab.

* The participants will sign consent forms and three casts will be taken on the first visit.
* The second visit will consist of fitting test socket A, which includes socket adjustments and the dynamic alignment. Once the socket is properly fit on the subject, we will begin their three trials (with two to three minute breaks in between trials) of the Time Up and Go assessment (TUG) followed by the Prosthesis Evaluation Questionnaire (PEQ) survey.
* Visit three will be comprised of socket B fitting, alignment, and testing. The subjects will proceed with the same procedure as stated in visit two. Following the outcome measures, participants will take the PEQ survey for socket B.
* Visit four is the final visit of testing and data collection. Socket C will be presented to the subject and they will go through the same dynamic alignment process and outcome testing as the previous visits. Once finished, the subjects will take the final PEQ survey on socket C and receive their compensation.

ELIGIBILITY:
Inclusion Criteria:

* K3-K4 level ambulator (Participants assessed as a K3 level are community ambulators, with the ability to tread on low level barriers and ambulate at variable speed. The highest K-level, (K4), is for high active, athletic ambulators with the ability or potential to ambulate at high impact, stress, or energy levels.)
* 18 years or older
* unilateral trans-tibial amputees with intact skin
* must have worn their prosthesis for at least 5 months

Exclusion Criteria:

* patients requiring a custom liner
* those on dialysis or have heart conditions
* patients requiring an assistive device (Examples of assistive devices would include; canes, walkers, forearm crutches, wheelchairs, hemi walkers, or rollators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | change between visit 1(baseline/start of study) and visit 2 (about 1 week fter visit 1)
  This assessment requires a standard armchair, a stopwatch, and a walkway clearly marked at 10 feet. The participant will be instructed to begin to walk on the word "Go". Promptly, the participant will stand up from the armchair, walk to the line on the floor at a normal pace, turn, then walk back to chair at their selected pace, and sit down again. Due to the fact that the participant will have to do this task three time they will be given a two to three minute resting period in between trials.

SECONDARY OUTCOMES:
Timed Up and Go Test | change between visit 1(baseline/start of study) and visit 3 (about 2 weeks after visit 1)
  This assessment requires a standard armchair, a stopwatch, and a walkway clearly marked at 10 feet. The participant will be instructed to begin to walk on the word "Go". Promptly, the participant will stand up from the armchair, walk to the line on the floor at a normal pace, turn, then walk back to chair at their selected pace, and sit down again. Due to the fact that the participant will have to do this task three time they will be given a two to three minute resting period in between trials.
Prosthesis Evaluation Questionnaire | change between visit 1(baseline/start of study) and visit 2 (about 1 week after visit 1)
  This questionnaire asks questions regarding the participant's socket, specific bodily sensations, pain in the residual limb, as well as social and emotional aspects of using a prosthesis.
Prosthesis Evaluation Questionnaire | change between visit 1(baseline/start of study) and visit 3 (about 2 weeks after visit 1)
  This questionnaire asks questions regarding the participant's socket, specific bodily sensations, pain in the residual limb, as well as social and emotional aspects of using a prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, MPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States